CLINICAL TRIAL: NCT01127646
Title: Assessing the Effect of Missing Doses (Off-Days) of Daily Medication in Patients Stable on Pharmacotherapy for ADHD Receiving Atomoxetine or OROS Methylphenidate: A Parallel Matched Group Clinical Study (On/Off Study)
Brief Title: A Study in Attention Deficit Hyperactivity Disorder in Children and Adolescents
Acronym: EMD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to lack of availability of study participants to accommodate the study design
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13070; B4Z-EW-LYEN (Other: Eli Lilly and Company); 2009-011426-33 (EudraCT Number)
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Results first posted 2012-06-04 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine (Experimental): Participants received 25-80 milligrams (mg) of atomoxetine orally, once daily during the run-in period for up to 7 days. The run-in period was followed by the 4-week on/off period in which participants received 25-80 mg of atomoxetine orally, once daily for 4 weeks, except for the off-days, where participants received 1 or 2 oral once daily placebo doses per week, with 6 nonconsecutive, double-blinded placebo doses in total over the 4-week on/off period. The on/off period was followed by a run-out period in which participants received 25-80 mg of atomoxetine orally, once daily for 1-5 days.
  Interventions: Drug: Atomoxetine; Drug: Placebo
- Osmotic-release oral system methylphenidate (Active Comparator): Participants received 18-54 mg of osmotic-release oral system (OROS) methylphenidate orally, once daily during the run-in period for up to 7 days. The run-in period was followed by the 4-week on/off period in which participants received 18-54 mg of OROS methylphenidate orally, once daily for 4 weeks, except for the off-days, where participants received 1 or 2 oral once daily placebo doses per week, with 6 nonconsecutive, double-blinded placebo doses in total over the 4-week on/off period. The on/off period was followed by a run-out period in which participants received 18-54 mg of OROS methylphenidate orally, once daily for 1-5 days.
  Interventions: Drug: Osmotic-release oral system methylphenidate; Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — 25-80 milligrams (mg) administered orally, once daily.
  Other Names: Strattera; LY139603
  Arms: Atomoxetine
Drug: Osmotic-release oral system methylphenidate — 18-54 mg administered orally, once daily.
  Arms: Osmotic-release oral system methylphenidate
Drug: Placebo — Administered orally, once daily for random nonconsecutive 6 days during 4-week treatment period.

SUMMARY:
The main purpose of the study is to help to understand the effect on children and adolescents who are stable on treatment with atomoxetine or osmotic-release oral system (OROS) methylphenidate for attention-deficit/hyperactivity disorder (ADHD) of not taking the medication for a maximum of 6 days over a 28-day study treatment period.

DETAILED DESCRIPTION:
The present study is designed to assess the effect of missed doses of daily medication (off-days). On the off-days the patient will take a placebo (sugar pill). Over the 4 weeks of the actual study there will be 6 random off-days of study medicine and neither the caregiver, patient nor study doctor will know which days are the missing days.

To cover all aspects of the patients' lives and notably their school time, aside from investigator's assessments, evaluations will also be performed on a daily basis by those involved in their day-to-day life: parents, teachers (on school days) and the patients themselves, using an electronic diary.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the Diagnostic and Statistical Manual for Mental Disorders, Fourth Edition Text Revision (DSM-IV-TR) diagnostic criteria for attention-deficit/hyperactivity disorder (ADHD), confirmed at screening by administering the Kiddie Schedule for Affective Disorders and Schizophrenia for School Aged Children-Present and Lifetime Version.
* Patients must have an Attention-Deficit/Hyperactivity Disorder Rating Scale - IV - Parent Version: Investigator Administered and Scored, total score of less than or equal to 20 at screening and baseline.
* Patients must have a Clinical Global Impression-Attention-Deficit/Hyperactivity Disorder-Improvement score of 1 ("very much better") or 2 ("much better") at screening and baseline.
* Patients must have been taking either atomoxetine or osmotic-release oral system methylphenidate for the treatment of ADHD between 3 and a maximum of 15 months prior to screening.
* Patients must have been receiving the same dose of atomoxetine or osmotic-release oral system methylphenidate as monotherapy in a single daily dose during the 4 weeks prior to screening.
* For females of child-bearing potential only: Test negative for pregnancy at the time of entry based on a urine pregnancy test
* Signed informed consent document (ICD)

Exclusion Criteria:

* Patients who weigh less than 20 kilograms (kg) or more than 70 kg at study entry
* Documented history of bipolar disorder, any history of psychosis or pervasive development disorder.
* Patients with a history of any seizure disorder or patients who have taken anticonvulsant treatment for seizure control.
* Patients at serious suicidal risk.
* History of severe allergies to more than one class of medications or have had multiple adverse drug reactions.
* Patients with acute or unstable medical conditions including cardiovascular disease and hypertension.
* Patients taking excluded concomitant medications or likely to begin structured psychotherapy for ADHD.
* Patients who are currently enrolled in, or discontinued within the last 30 days from a clinical trial.
* Sexually active females who do not use a medically acceptable method of contraception.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- Netherlands (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arnhem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Capelle aan den IJssel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maastricht
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donostia / San Sebastian
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Esplugues de Llobregat
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
- Sweden (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gothenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Handen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uppsala

RESULTS

PARTICIPANT FLOW:
Groups:
- Atomoxetine: Participants received 25-80 milligrams (mg) of atomoxetine orally, once daily for 4 weeks (on/off period), except for the off-days, where participants received 1 or 2 oral once daily placebo doses per week, with 6 nonconsecutive, double-blinded placebo doses in total over the 4-week on/off period.
- Osmotic-Release Oral System (OROS) Methylphenidate: Participants received 18-54 mg of OROS methylphenidate orally, once daily for 4 weeks (on/off period), except for the off-days, where participants received 1 or 2 oral once daily placebo doses per week, with 6 nonconsecutive, double-blinded placebo doses in total over the 4-week on/off period.
Period: Overall Study
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Started | 15 | 8
Completed | 14 | 7
Not Completed | 1 | 1
Not completed — Entry Criteria Not Met | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate | Total
Number analyzed (Participants) | 15 | 8 | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 10.8 (2.65) | 10.9 (2.80) | 10.8 (2.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 12 | 6 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 7 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 1 | 0 | 1
  Spain | 12 | 8 | 20
  Sweden | 2 | 0 | 2
Attention-Deficit/Hyperactivity Disorder (ADHD) Subtype: Current Episode [Number; unit: participants]
  Combined | 7 | 4 | 11
  Hyperactive/Impulsive | 0 | 1 | 1
  Inattentive | 1 | 0 | 1
  Subtype not present | 6 | 3 | 9
  Missing | 1 | 0 | 1
Attention-Deficit/Hyperactivity Disorder (ADHD) Subtype: Lifetime Episode [Number; unit: participants] — Lifetime episode refers to the most severe episode in the past.
  participants
    Combined | 8 | 7 | 15
    Hyperactive/Impulsive | 0 | 1 | 1
    Inattentive | 5 | 0 | 5
    Subtype not present | 1 | 0 | 1
    Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Daily Parent Report of Evening and Morning Behavior-Revised (DPREMB-R) Scale Mean Total Score (On-Days Versus Off-Days) During the 4-Week Treatment Period
Description: Parent-completed 11-item questionnaire; measures difficulty level of and 8 common evening behaviors (such as, sit through dinner) and 3 common morning behaviors (such as, get out of bed). Each item is scored on a 4-point Likert scale ranging from 0 (no difficulty) to 3 (a lot of difficulty). Total score (evening+morning) range is 0 to 33. Higher scores indicate greater difficulty in evening and morning behavior. DPREMB-R total score between days without missing doses (on-days) and days with missing doses (off-days) was not analyzed due to the insufficient sample size.
Time Frame: Baseline through 4 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Global Impression of Perceived Difficulties (GIPD) Scale-Patient Version Total Score and Individual Items (On-Days Versus Off-Days) During the 4-Week Treatment Period
Description: Assesses attention-deficit/hyperactivity disorder (ADHD)-related difficulties (overall difficulties perceived in morning, during school, during homework, in evening, over entire day and night). Participant rates difficulties during past week on 7-point scale (1=normal, not difficult at all; 7=extremely difficult) for each of 5 items. Total score=sum of all subscores (items); range: 5 to 35. Higher scores=greater impairment. GIPD-Pat total score and item scores between days without missing doses (on-days) and days with missing doses (off-days) were not analyzed due to insufficient sample size.
Time Frame: Baseline through 4 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Conners' Global Index-Teacher Rating Scale Total Score (On-Days Versus Off-Days) During the 4-Week Treatment Period
Description: The teacher version of Conners' Global Index consists of 10 items with each item being scored on a 4-point scale ranging from 0 (not true at all, or never/seldom) to 3 (very much true, or very often/very frequent). The total score ranges from 0 to 30. Higher scores indicate greater impairment. The Conner's Global Index-Teacher Rating Scale total score between days without missing doses (on-days) and days with missing doses (off-days) was not analyzed due to the insufficient sample size.
Time Frame: Baseline through 4 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Global Impression of Perceived Difficulties Scale-Patient Version (GIPD-Pat) Scale Total Score and Individual Items During the 4-Week Treatment Period
Description: Assesses attention-deficit/hyperactivity disorder (ADHD)-related difficulties (overall difficulties perceived in morning, during school, during homework, in evening, over entire day and night). Difficulties during past week are rated by participant on a 7-point scale (1=normal, not difficult at all; 7=extremely difficult) for each of 5 items. Total score=sum of all subscores (items); range: 5 to 35. Higher scores=greater impairment. Mean GIPD-Pat total score and individual item scores for days with missing doses (off-days) between both groups were not analyzed due to insufficient sample size.
Time Frame: Baseline through 4 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Attention-Deficit/Hyperactivity Disorder Rating Scale-Parent Version: Investigator Administered and Scored (ADHD-RS-IV Parent:Inv) Total Score and Subscores at Weeks 2, 3, and 4
Description: Assesses 18 Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) ADHD diagnosis symptoms/severity in past week. Each item: 0 (none/never, rarely) to 3 (severe/very often). Total score ranges from 0 to 54. Higher total scores indicate greater illness severity. This outcome measure was not analyzed due to the insufficient sample size.
Time Frame: Weeks 2, 3, and 4
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Clinical Global Impression-Attention Deficit/Hyperactivity Disorder-Severity Scale (CGI-ADHD-S) at Weeks 2, 3, and 4
Description: This instrument is a single-item expert rating of the severity of the participant's attention-deficit/hyperactivity disorder (ADHD) symptoms in relation to the assessor's total experience of participants with ADHD. Severity is rated on a 7-point scale (1=normal, not ill at all; 7=among the most extremely ill participants). Higher scores represent greater illness severity. This outcome measure was not analyzed due to the insufficient sample size.
Time Frame: Weeks 2, 3, and 4
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Emotion Expression Scale for Children (EESC)-Parent Rated Total Score up to Week 5
Description: 29-item parent-reported measure used to monitor effect of attention-deficit/hyperactivity disorder (ADHD) medication; examines 3 aspects of emotion expression: positive emotions, emotional flatness, and emotional lability. Each item rated on 5-point Likert scale (1="not at all true" to 5="very much true"). Positive emotional subscale items reversed scored (6-raw score). Total score=transformed positive emotion + emotional flatness+ emotional lability subscales. Total scores range: 29 to 145. Higher scores=emotional impairment. This outcome measure not analyzed due to insufficient sample size.
Time Frame: Up to Week 5
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Groups:
- Atomoxetine: Participants received 25-80 milligrams (mg) of atomoxetine orally, once daily for 4 weeks (on/off period), except for the off-days, where participants received 1 or 2 oral once daily placebo doses per week, with 6 nonconsecutive, double-blinded placebo doses in total over the 4-week on/off period. The on/off period was followed by a run-out period in which participants received 25-80 mg of atomoxetine orally, once daily for 1-5 days.
- Osmotic-Release Oral System (OROS) Methylphenidate: Participants received 18-54 mg of OROS methylphenidate orally, once daily for 4 weeks (on/off period), except for the off-days, where participants received 1 or 2 oral once daily placebo doses per week, with 6 nonconsecutive, double-blinded placebo doses in total over the 4-week on/off period. The on/off period was followed by a run-out period in which participants received 18-54 mg of OROS methylphenidate orally, once daily for 1-5 days.
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Daily Parent Report of Evening and Morning Behavior-Revised (DPREMB-R) Scale Subscores (On-Days Versus Off-Days) During the 4-Week Treatment Period
Description: Parent-completed 11-item questionnaire; measures difficulty level of 8 common evening behaviors (such as, sit through dinner) and 3 common morning behaviors (such as, get out of bed) from 0 (no difficulty) to 3 (a lot of difficulty). Evening behavior total score range is 0 to 24. Morning behavior total score range is 0 to 9. Higher scores indicate greater difficulty in evening and morning behavior. DPREMB-R subscores between days without missing doses (on-days) and days with missing doses (off-days) not analyzed due to insufficient sample size.
Time Frame: Baseline through 4 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Patient Outcomes Questions (On-Days Versus Off-Days) During the 4-Week Treatment Period
Description: 6-item questionnaire from attention-deficit/hyperactivity disorder (ADHD) advocacy group evaluates treatment outcomes ADHD participant's perspective. Parent completed on each day of on/off period. Each item ranged from 1 ("I totally agree") to 5 ("I totally disagree"). Items 1 and 2 pertain to sleeping and eating; high scores=better outcome. Items 3-6 pertain to behavior; high scores=worse outcome. The mean scores for analysis would have been created for each question across the days of each of the on and off phases; however, mean scores were not analyzed due to insufficient sample size.
Time Frame: Baseline through 4 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Daily Parent Report of Evening and Morning Behavior-Revised (DPREMB-R) Scale Total Score and Subscores During the 4-Week Treatment Period
Description: Parent-completed 11-item questionnaire; measures difficulty level of 3 common morning behaviors (such as, get out of bed) and 8 common evening behaviors (such as, sit through dinner) from 0 (no difficulty) to 3 (a lot of difficulty). Evening behavior total score range is 0 to 24. Morning behavior total score range is 0 to 9. Total score (evening+morning) range is 0 to 33. Higher scores indicate greater difficulty in evening and morning behavior. Mean DPREMB-R total score and subscores for days with missing doses (off-days) between both groups were not analyzed due to insufficient sample size.
Time Frame: Baseline through 4 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Conners' Global Index-Teacher Rating Scale Total Score During the 4-Week Treatment Period
Description: The teacher version of Conners' Global Index consists of 10 items with each item being scored on a 4-point scale ranging from 0 (not true at all, or never/seldom) to 3 (very much true, or very often/very frequent). The total score ranges from 0 to 30. Higher scores indicate greater impairment. The Conners' Global Index-Teacher Rating Scale total score for days with missing doses (off-days) between both groups were not analyzed due to insufficient sample size.
Time Frame: Baseline through 4 weeks
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Global Impression of Perceived Difficulties Investigator Version (GIPD-Inv) Total Score and Subscores At Weeks 2, 3, and 4
Description: Assesses attention-deficit/hyperactivity disorder (ADHD)-related difficulties (overall difficulties perceived in morning, during school, during homework, in evening, and over entire day and night). Difficulties during past week are rated by investigator on a 7-point scale (1=normal, not difficult at all; 7=extremely difficult) for each of 5 items. Total score=sum of all subscores (items) and ranges from 5 to 35. Higher scores indicate greater impairment. This outcome measure was not analyzed due to the insufficient sample size.
Time Frame: Weeks 2, 3, and 4
Population: No participants had data analyzed due to the termination of the trial and the insufficient sample size.
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Change From Baseline in Heart Rate up to 5 Weeks
Time Frame: Baseline, up to 5 weeks
Population: Safety population: all participants who entered the study and took at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Number analyzed (Participants) | 14 | 7
beats per minute (bpm) | -1.2 (7.65) | 2.5 (12.74)

14. Other Pre Specified Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure up to 5 Weeks
Time Frame: Baseline, up to 5 weeks
Population: Safety population: all participants who entered the study and took at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Number analyzed (Participants) | 14 | 7
millimeters of mercury (mm Hg)
  Diastolic Blood Pressure | 1.9 (6.14) | -1.5 (4.67)
  Systolic Blood Pressure | -0.1 (9.00) | -3.7 (3.75)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the entire study period, which included the following: 3-14 day screening period, a run-in period of up to 7 days, a 4-week on/off period, and a 1-5 day run-out period for a maximum of 54 days.
Groups:
- Osmotic-Release Oral System (OROS) Methylphenidate: Participants received 18-54 mg of OROS methylphenidate orally, once daily during the run-in period for up to 7 days. The run-in period was followed by the 4-week on/off period in which participants received 18-54 mg of OROS methylphenidate orally, once daily for 4 weeks, except for the off-days, where participants received 1 or 2 oral once daily placebo doses per week, with 6 nonconsecutive, double-blinded placebo doses in total over the 4-week on/off period. The on/off period was followed by a run-out period in which participants received 18-54 mg of OROS methylphenidate orally, once daily for 1-5 days.
Arm/Group | Atomoxetine | Osmotic-Release Oral System (OROS) Methylphenidate
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/8
Other Adverse Events (participants affected / at risk) | 7/15 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=15) | Osmotic-Release Oral System (OROS) Methylphenidate (N=8)
Abdominal pain (Gastrointestinal disorders) | 1 (6) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (10) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (8) | 0 (0)
Somnolence (Nervous system disorders) | 1 (3) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0)
Impulsive behaviour (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study (Study LYEN) was terminated after enrolling 23 participants due to lack of availability of study participants to accommodate the study design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days